CLINICAL TRIAL: NCT04850131
Title: Mesh Free Desarda Repair Compared With Lichtenstein Repair for the Treatment of Primary Inguinal Hernias
Brief Title: Desarda Repair Compared to Lichtenstein Repair for the Treatment of Inguinal Hernias
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benazir Bhutto Hospital, Rawalpindi (Other Government)
Responsible Party: Principal Investigator, Muhammad Usman Ghani, SENIOR REGISTRAR SURGERY, Benazir Bhutto Hospital, Rawalpindi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 274/IREF\RMU\2020
Record Dates: First submitted 2021-04-10; First posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Postoperative Pain; Recurrence; Wound Complication
Keywords: Desarda Repair; Comparison; Lichtenstein Repair; Randomized Controlled Trial
MeSH Terms: conditions — Pain, Postoperative; Recurrence

STUDY DESIGN:
Intervention Model Description: A total of 82 patients with inguinal hernias were selected randomly to participate in this study. They were subjected to either Lichtenstein hernioplasty or Desarda herniorrhaphy. A follow-up was conducted to analyze the hospital stay, return to work, recurrence rate, chronic pain, postoperative complications, and cost-effectiveness.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Desarda (Active Comparator): Forty-one patients who were randomly assigned to the Desarda group underwent the Desarda repair for their problem. Patients were followed for various data point values during operation, immediately after the operation, and for a period of one year post-operatively.
  Interventions: Procedure: Desarda repair
- Lichtenstein (Active Comparator): Forty-one patients randomly assigned to the Lichtenstein group underwent the standard mesh repair and were followed for the same data point values and variables for the same specified period of time.
  Interventions: Procedure: Desarda repair

INTERVENTIONS:
Procedure: Desarda repair — Desarda is a new tissue-based technique developed from applying the externally oblique muscle aponeurosis in the form of an undetached strip making the posterior wall in the inguinal canal stiffer. This paper focuses on analyzing comparisons between mesh-free Desarda repair and the Lichtenstein technique for the treatment of hernia inguinalis
  Other Names: Lichtenstein repair

SUMMARY:
The Lichtenstein technique for hernia repair is safe and simple, but the underlying mesh prosthesis has its setbacks, as it acts as a mechanical barrier5. The mesh does not provide mobile and the physiologically dynamic posterior wall. The most dangerous complication associated with the mesh prosthesis is its migration from the abdominal cavity's primary implantation site. The relatively knew technique developed by Dr. Desarda does not utilize the synthetic mesh rather it uses a strip of external oblique aponeurosis to strengthen the posterior wall. Our study has compared the two methods regarding various aspects.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of age between 20 to 70years
2. A primary inguinal hernia
3. Consented to participate in the research.

Exclusion Criteria:

1. Age below 20,
2. Recurrent and pantaloons hernia
3. Patients who did not give the informed consent
4. Patients who lose the follow-up

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 24 hours after the surgery
  Measured on Visual analogue scale (VAS) where 0 meaning no pain and 10 means worst pain
Postoperative pain | 3 months after the primary surgery
  Measured on Visual analogue scale (VAS) where 0 meaning no pain and 10 means worst pain
Recurrence | Within 01 year of the primary surgery
  Described as reappearance of the inguinal hernia on the operated side

SECONDARY OUTCOMES:
Wound complication | Complications occuring within 30 days after the surgery
  Described as number of patients developing the wound complications like seroma , hematoma formation and surgical site infection.

CONTACTS AND LOCATIONS:
Overall Officials: MUHAMMAD USMAN GHANI, FCPS, Principal Investigator — BENAZIR BHUTTO HOSPITAL
Locations (1):
- Benazir Bhutto Hospital Rawalpindi, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No